CLINICAL TRIAL: NCT03464305
Title: A Phase III Double-blind Placebo-controlled Randomised Trial of Aspirin on Recurrence and Survival in Colon Cancer Patients
Brief Title: ASPIRIN Trial Belgium
Acronym: ASPIRIN
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: University Hospital, Antwerp (Other)
Collaborators: Kom Op Tegen Kanker (Other); Anticancerfund (Unknown)
Responsible Party: Principal Investigator, ethisch.comite@uza.be, Prof. dr. Marc Peeters, Diensthoofd Oncologie, University Hospital, Antwerp
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: BE 2017-001397-41
Record Dates: First submitted 2018-03-07; First posted 2018-03-14 (Actual); Last update posted 2024-03-19 (Actual); Status verified 2024-03

CONDITIONS: Colon Cancer
Keywords: Colonic Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Colonic Diseases; Aspirin; Recurrence; Digestive System Diseases; Intestinal Diseases; Disease Attributes; Pathologic Processes
MeSH Terms: conditions — Colonic Neoplasms; Colorectal Neoplasms; Intestinal Neoplasms; Gastrointestinal Neoplasms; Digestive System Neoplasms; Neoplasms by Site; Neoplasms; Colonic Diseases; Recurrence; Digestive System Diseases; Intestinal Diseases; Disease Attributes; Pathologic Processes | interventions — Aspirin

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aspirin (Experimental): Patients treated with acetylsalicylic acid 80 mg once daily for 5 years. Patients will be stratified according to the admission of adjuvant chemotherapy.
  Interventions: Drug: acetylsalicylic acid
- Placebo (Placebo Comparator): Patients treated with placebo. Patients will be stratified according to the admission of adjuvant chemotherapy.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: acetylsalicylic acid — Patients treated with acetylsalicylic acid 80 mg once daily for 5 years. Patients will be stratified according to the admission of adjuvant chemotherapy.
  Arms: Aspirin
Drug: Placebo — Patients treated with placebo. Patients will be stratified according to the admission of adjuvant chemotherapy.
  Arms: Placebo

SUMMARY:
The purpose of this study is to determine whether acetylsalicylic acid is effective on the recurrence and survival of colon cancer patients.

DETAILED DESCRIPTION:
The purpose of this study is to determine the effect of 80mg acetylsalicylic acid (given orally once daily for 5 years) on 5 year overall survival (OS) for stage II and III colon cancer patients of 45 years of age and older. Preclinical, epidemiologic and clinical evidence suggest that acetylsalicylic acid use may reduce overall cancer risk and mortality in colon cancer patients. It is a phase III double blind placebo controlled, randomized trial of adjuvant low-dose acetylsalicylic acid in colon cancer patients. Patients will be stratified at randomization by centre, age (<70 and ≥70 years) chemotherapy use (any versus none) and disease stage.

ELIGIBILITY:
Inclusion Criteria:

* Patients 45 years and older with histologically confirmed adenocarcinoma of the colon
* Patients must have TNM stage that is one of the following: pT3-4; N0-2 and M0, or pT1-2 and N1-2 (Union for International Cancer Control (UICC) stage II and III) (in case of >1 tumour: more advanced tumour is stage II or III)
* Patients must have completed surgical resection (R0) (both laparoscopic and open surgery) within 12 weeks of randomization

Exclusion Criteria:

* Patients with rectal cancer (defined as tumour within 15 cm from the anal verge)
* Patients currently taking oral anti-coagulants or use of LMWH or use of DOACs
* Patients currently taking (low-dose) acetylsalicylic acid or other anti-aggregantia for any reason
* Patients with a history of bleeding disorders or active gastric or duodenal ulcers
* Patients currently taking high dose systemic glucocorticoids (≥ 30 mg predniso(lo)n or equivalent)
* Patients with (suspected) (non-) polyposis syndrome (FAP/AFAP, MAP, Lynch syndrome)
* Patients with >100 polyps of the colon or a known hereditary syndrome of the colon in a first degree family member
* Allergy or intolerance to salicylates
* Patients with local or distant recurrent disease
* Previous malignancies other than CIN or SCC with a disease free survival less than 5 years
* Presence of any psychological, familial, sociological or geographical condition potentially hampering compliance with the study protocol and follow-up schedule; those conditions should be discussed with the patient before registration in the trial

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 148 (Actual)
Dates: Start 2018-02-22 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
5 year overall survival | 5 years
  The time to an event for OS is defined as the time interval between the date of randomisation and the date of death.

SECONDARY OUTCOMES:
Disease Free Survival | 5 years
  The time to an event for DFS is defined as the time interval between the date of randomisation and the date of disease recurrence or death, whichever comes first. Recurrence of a disease can be a loco-regional recurrence, a distant recurrence or a new primary colon cancer. The evidence for recurrence must be documented in the patients' file.
Time to Treatment Failure | 5 years
  The time elapsed between randomisation until treatment discontinuation due to disease progression, unacceptable toxicity, death or any other event of interest.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Peeters, Prof dr, Principal Investigator — University Hospital, Antwerp
Locations (29):
- Belgium (29):
  - AZ Rivierenland campus Bornem (Sint Jozefkliniek), Bornem, Antwerpen
  - AZ Klina, Brasschaat, Antwerpen
  - AZ Monica, Deurne, Antwerpen
  - UZ Antwerpen, Edegem, Antwerpen
  - AZ Rivierenland campus Rumst (Heilige Familie), Rumst, Antwerpen
  - VITAZ (AZ Nikolaas), Sint-Niklaas, Oost-Vlaanderen
  - Ziekenhuis Netwerk Antwerpen (ZNA), Antwerp
  - Gasthuiszusters Ziekenhuizen (GZA), Antwerp
  - Clinique Saint-Luc, Bouge
  - AZ Sint-Lucas, Bruges
  - CHIREC, Brussels
  - Grand Hôpital de Charleroi, Charleroi
  - AZ Sint-Blasius, Dendermonde
  - AZ Alma, Eeklo
  - AZ Sint-Dimpna, Geel
  - AZ Maria Middelares, Ghent
  - Jessa Ziekenhuis, Hasselt
  - AZ Groeninge, Kortrijk
  - RZ Heilig Hart, Leuven
  - CH de l'Ardenne, Libramont
  - CHR de la Citadelle, Liège
  - CHU Ambroise Paré, Mons
  - CH de Mouscron, Mouscron
  - CHU UCL Namur Site de Sainte-Elisabeth, Namur
  - Clinique Saint-Pierre, Ottignies-Louvain-la-Neuve
  - AZ Glorieux, Ronse
  - AZ Sint-Trudo, Sint-Truiden
  - CHR Verviers, Verviers
  - OLV van Lourdes Ziekenhuis, Waregem

REFERENCES:
- See also: Aspirin Trialist Collaborative Group — https://www.lumc.nl/org/atcg/participating-trials/ASPIRINBE/

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2020-03-26): https://cdn.clinicaltrials.gov/large-docs/05/NCT03464305/Prot_SAP_000.pdf